CLINICAL TRIAL: NCT04936191
Title: Dynamic Change of Coronary Artery Curvature After Adaptive Remodeling
Brief Title: Dynamic Change of Coronary Artery Curvature
Acronym: DC3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202101142DIPA
Record Dates: First submitted 2021-05-30; First posted 2021-06-23 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Drug eluting stent; Coronary intervention; Coronal curvature
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DynamX Bioadaptor (Experimental): Patients were randomized during the percutaneous coronary intervention before stent implantation and assigned to the study arm using an electronic spreadsheet indicating the group assignment by random numbers. The patients will be 1:1 randomized to 2 groups: DynamX Bioadaptor and DESyne DES groups.
  Interventions: Device: DynamX Bioadaptor
- DESyne Drug-eluting Stent (Active Comparator): Patients were randomized during the percutaneous coronary intervention before stent implantation and assigned to the study arm using an electronic spreadsheet indicating the group assignment by random numbers. The patients will be 1:1 randomized to 2 groups: DynamX Bioadaptor and DESyne DES groups.
  Interventions: Device: DynamX Bioadaptor

INTERVENTIONS:
Device: DynamX Bioadaptor — Patients received percutaneous coronary intervention in a similar way to a traditional DES. Patients first receive radial artery or femoral artery cannulation with anticoagulation during the intervention. All coronary angiograms are carefully measured by at least 2 orthographic views and performed under the same standard conditions. After adequate predilatation of the target lesion, the coronary stenting will be performed. All patients will receive a loading dose of acetylsalicylic acid and a P2Y12 inhibitor pre-procedure followed by dual antiplatelet therapy for at least 6 months.
  Other Names: DESyne Drug-eluting Stent

SUMMARY:
The novolimus-eluting DynamX bioadaptor system is composed of 71 µm cobalt-chromium sinusoidal rings connected to each other axially by three S-links Each ring contains three uncaging elements that are positioned at equal distance in low stress regions of struts oriented in a helical configuration along the length of the bioadaptor which remain intact after uncaging. The uncaging elements consist of three separable junctions per ring held together by a 6 µm polymer coating that is resorbed over six months, allowing uncaging of the vessel and adaptive remodeling. Previous study showed the DynamX biodaptor is safe and effective treating in de novo coronary lesion. It also increased of vessel and device area while maintain in the mean lumen area after one year follow-up. However, the unchanging effect of Dynamx bioadaptor on coronary geometry change remained unknown. The present randomized control study is designed to investigate the differences of dynamic coronary artery geometry changes evaluated by coronary computed tomography angiography after DynamX Bioadaptor and permanent metallic DES implantation.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the most common type of heart disease and the leading cause of death worldwide. Percutaneous coronary intervention and coronary artery bypass graft are the guideline suggested treatment. Drug-eluting stents (DES) is the guideline suggested treatment options. Percutaneous coronary intervention with DES provides not just acute luminal gains, but also good long-term patency and clinical outcomes. However, in-stent neoatherosclerosis, very late stent thrombosis, and endothelial dysfunction remained important long-term issues. In addition, metallic stent encages the vessel segment, limits its remodeling and vasomotor function. The original vessel geometry, curvature, tortuosity, and wall shear stress, which are associated with plaque formation are also changed permanently by stent implantation. Although bioresorbable scaffolds attempted to address these issues by providing structural support to the vessel early on, followed by resorption, randomized trials showed that, prior to their resorption, they were less safe and effective than contemporary DES. Since that, the novel DES, DynamX Bioadaptor, is designed to improve these limitations.

The novel DES, DynamX Bioadaptor, is designed to restore normal pulsatility and adaptive remodeling in blood vessels after stent implantation. It is a cobalt-chromium stent with a biodegradable polymer coating that releases novolimus. Segments of the stent are held together by the polymer coating, which is designed to be fully absorbed in 6 months. After degradation of polymer, the stent struts unlink and uncage the stented segment. Pilot study demonstrated vessel uncaging and restoration of cyclic pulsatility 12 months after DynamX Bioadaptor implantation. Adaptive remodeling 12 months after DynamX Bioadaptor implantation will restore flexibility and natural geometry of the stented vessel segment. Thus, the dynamic beat-to-beat (cardiac cycle) changes of curvature and tortuosity will be more pronounced in the DynamX Bioadaptor group compared with that in the permanent metallic Elixir DESyne DES group. The DynamX Bioadaptor can potentially restore the vessel geometry and improve outcomes. The present randomized control study is designed to investigate the differences of dynamic coronary artery geometry changes after DynamX Bioadaptor and permanent metallic DES implantation, using coronary computed tomography angiography (CCTA) as an evaluation tool.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 20 years old.
* Written informed consent can be obtained.
* The enrolled coronary vessel only has one target coronary lesion required stenting.
* The target coronary lesion is 50 to 100% stenosis and stenting is required.
* Coronary artery de novo lesion requiring implantation of a single drug eluting stent with length ≥ 32 mm.
* Patients are able to tolerate dual antiplatelets for at least six months.

Exclusion Criteria:

* Patient is unwilling to join this study.
* Patients have end-stage renal disease under dialysis, chronic kidney disease (serum creatine > 1.5 mg/dL), symptomatic heart failure, active cancer, high bleeding risk, ST elevation myocardial infarction or hemodynamic unstable non-ST elevation myocardial infarction.
* Coronary lesion with following features: heavily calcification, ostial lesion, lesions requiring post-stenting side branch dilatation and lesions required more than one stent to treat.
* The left ventricular ejection fraction is ≤ 40%.
* No scheduled operation within six months after the coronary stenting is allowed unless continuous dual antiplatelet use is acceptable.
* Patients are unsuitable or unable to receive CCTA.
* Pregnant women or women with breast feeding or suitable pregnant women without contraception during the study period.
* Patient is currently participating another interventional trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The differences of vessel geometry | 12 months ± 2 weeks
  The differences of vessel geometry during systolic-diastolic phases, 12 months ± 2 weeks after DynamX Bioadaptor or Elixir DESyne DES implantation, measured by CCTA.

SECONDARY OUTCOMES:
New plaque formation related in-stent/in-segment restenosis | 12 months ± 2 weeks
  In-stent/in-segment restenosis 12 months ± 2 weeks after DynamX Bioadaptor or Elixir DESyne DES implantation, measured by CCTA.

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Li Kao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Cheng-Hsuan Tsai, Taipei, Please Select:, Taiwan

IPD SHARING:
Plan to Share IPD: No
The IPD data only could be shared after discuss with the principle investigator.

REFERENCES:
- [Result] Verheye S, Vrolix M, Montorfano M, Zivelonghi C, Giannini F, Bedogni F, Dubois C, De Bruyne B, Costa RA, Chamie D, de Ribamar Costa J Jr, Kereiakes DJ, Abizaid AA, Colombo A. Twelve-month clinical and imaging outcomes of the uncaging coronary DynamX bioadaptor system. EuroIntervention. 2020 Dec 18;16(12):e974-e981. doi: 10.4244/EIJ-D-20-00763. PMID 32894231
- [Derived] Tsai CH, Chu HH, Huang CC, Yeh CF, Chen YH, Lin MS, Ko TY, Chen CK, Huang YC, Chiang PY, Lee WJ, Kao HL. Dynamic Change of Coronary Artery Geometry After Bioadaptor Implantation: A Single-blind Randomized Controlled Trial. Circ Cardiovasc Interv. 2026 Jan 29:e016191. doi: 10.1161/CIRCINTERVENTIONS.125.016191. Online ahead of print. PMID 41608781